CLINICAL TRIAL: NCT07065058
Title: A Phase I, Single-Center, Open-Label, Single-Arm, Fixed-Sequence Clinical Study to Evaluate the Pharmacokinetic Interactions of VCT220 With Repaglinide, Rosuvastatin, and Digoxin in Healthy, Overweight, and Obese Subjects
Brief Title: A Drug Drug Interaction Study to Evaluate the Effect of VCT220 on the Pharmacokinetics of Repaglinide, Rosuvastatin, and Digoxin in Healthy, Overweight, and Obese Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VCT220-I-04-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — repaglinide; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): During the monotherapy phase, subjects receive repaglinide, rosuvastatin, and digoxin. After a 1-week washout period, VCT220 is administered starting from 20 mg and titrated up to 160 mg, followed by repeat administration of repaglinide, rosuvastatin, and digoxin.
  Interventions: Drug: Drug: VCT220, Repaglinide, Rosuvastatin, and Digoxin

INTERVENTIONS:
Drug: Drug: VCT220, Repaglinide, Rosuvastatin, and Digoxin — Single dose of Repaglinide at Day 2, Rosuvastatin and Digoxin at Day 3 Orally VCT220 once daily from Day 9 to Day 78, titrated from 20mg to 160mg. Co-administrated Repaglinide at Day 72, co-administrated Rosuvastatin and Digoxin at Day 73

SUMMARY:
This is a single-center, open-label, single-arm, fixed-sequence Phase I study in healthy, overweight, and obese subjects. The primary objective is to evaluate the effect of orally administered VCT220 tablets on the pharmacokinetics and safety of repaglinide , rosuvastatin, and digoxin.

A total of 24 subjects will be enrolled. Repaglinide is administered alone on Day 1 and coadministered with VCT220 on Day 72. Rosuvastatin and digoxin are administered together on Day 2 and again on Day 73 with VCT220. VCT220 will be titrated from 20 mg to 160 mg once daily from Day 9 to Day 78.

All study drugs are given under controlled fed or fasting conditions, with standardized water and meal restrictions. Intensive PK sampling will be conducted around dosing to assess any drug-drug interactions. Safety assessments will be conducted throughout the study.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm, fixed-sequence Phase I clinical study designed to evaluate the effect of orally administered VCT220 tablets on the pharmacokinetics (PK) and safety of repaglinide, rosuvastatin, and digoxin in healthy, overweight, and obese adult subjects. These three drugs are probe substrates for key drug transporters: repaglinide for OATP1B1/OATP1B3, rosuvastatin for BCRP, and digoxin for P-glycoprotein (P-gp).

A total of 24 subjects will be enrolled. On Day 1, subjects receive a single dose of repaglinide 0.5 mg under fasting conditions. On Day 2, rosuvastatin 10 mg and digoxin 0.25 mg are co-administered under fed conditions. From Day 9 to Day 78, subjects will receive VCT220 orally once daily after breakfast in an ascending dose regimen: 20 mg, 40 mg, 80 mg, 120 mg, and finally 160 mg, titrated every 2 weeks.

On Day 72, repaglinide is administered again under fasting conditions, now in the presence of steady-state VCT220. On Day 73, rosuvastatin and digoxin are administered again under fed conditions with VCT220. Water intake is restricted within 1 hour before and after dosing, and standardized meals are provided to control for food effects.

Serial blood samples will be collected before and after dosing for PK assessments. The primary endpoints are the PK parameters (Cmax, AUC) of the probe drugs with and without VCT220. Safety will be evaluated throughout the study via clinical assessments, laboratory tests, vital signs, ECGs, and adverse event monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be fully informed of the purpose, content, procedures, and potential adverse reactions of the study, voluntarily agree to participate, and sign the informed consent form (ICF) prior to any study-related procedures.
2. Male and female subjects aged between 18 and 65 years (inclusive).
3. Male subjects must weigh ≥50.0 kg and female subjects ≥45.0 kg, with a body mass index (BMI) ≥20 kg/m² [BMI = weight (kg) / height² (m²)].
4. Subjects must have no plans for childbearing from the time of signing the ICF until 3 months after the last dose of the study drug and must voluntarily agree to use effective contraception; subjects must also have no plans to donate sperm or eggs during this period.
5. Subjects must be able to communicate well with the investigators, and understand and comply with all study requirements.

Exclusion Criteria:

1. Any of the following laboratory abnormalities at screening:

   1. HbA1c ≥ 6.5%;
   2. Fasting plasma glucose (FPG) ≥ 7.0 mmol/L;
   3. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m² (calculated by CKD-EPI formula);
   4. ALT and/or AST > 1.5× upper limit of normal (ULN);
   5. Total bilirubin (TBIL) > 1.5× ULN;
   6. Serum amylase or lipase > 1.5× ULN;
   7. Calcitonin ≥ 1.0× ULN;
   8. Hemoglobin < 110 g/L (males) or < 100 g/L (females).
2. Positive test results for any of the following: HBsAg, HCV-Ab, HIV-Ab, or TP-Trust (syphilis).
3. 12-lead ECG during screening showing second- or third-degree atrioventricular block, long QT syndrome, QTcF ≥ 450 ms (males) or ≥ 470 ms (females) (QTcF = QT/RR^0.33), bundle branch block, Wolff-Parkinson-White syndrome, or other clinically significant arrhythmias (excluding sinus arrhythmia), or ECG findings deemed clinically significant by the investigator.
4. Known allergy to VCT220, repaglinide, rosuvastatin, or digoxin, or history of allergy to two or more drugs or foods.
5. Presence of clinically significant diseases requiring exclusion, including but not limited to disorders of the nervous, cardiovascular (unless deemed acceptable by the investigator), hematologic, lymphatic, immune, digestive, urinary, respiratory, metabolic, or skeletal systems.
6. History or current diagnosis of pancreatitis (acute or chronic), history of acute gallbladder disease (except for those who have undergone cholecystectomy), or clinically significant findings on baseline abdominal ultrasound.
7. Diagnosis of type 1, type 2, or other specific types of diabetes.
8. Use of GLP-1 receptor agonists within 6 months before screening.
9. Swallowing difficulties or gastrointestinal diseases affecting drug absorption (e.g., diarrhea, vomiting, IBD, acute gastroenteritis, peptic ulcer, or significant GI dysfunction with impaired absorption).
10. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
11. Major depressive disorder or other severe psychiatric disorders within 2 years prior to screening.
12. Surgery within 3 months prior to screening, planned surgery during the study, or history of surgeries that may affect ADME of drugs.
13. History of drug abuse or illicit drug use within 12 months prior to screening, or positive drug screen.
14. Participation in another drug/device trial within 3 months before screening or plans to participate in another clinical trial during the study.
15. Use of oral contraceptives within 30 days before screening (female subjects).
16. Use of long-acting estrogen or progestin injections, hormone-releasing IUDs, or implants within 6 months prior to screening (female subjects).
17. Blood donation (including components) or significant blood loss ≥400 mL, transfusion, or use of blood products within 3 months before screening.
18. Use of any prescription medications (especially those affecting CYP3A4, CYP2C8, CYP2C9, CYP2C19), over-the-counter drugs, herbal supplements, or dietary supplements within 14 days prior to first dosing, or plan to use them during the study.
19. Smoking more than 5 cigarettes per day within 3 months before screening, or inability to abstain from tobacco products during the study.
20. Alcohol consumption >14 units/week (1 unit ≈ 360 mL beer at 5% alcohol, 45 mL liquor at 40%, or 150 mL wine at 12%) within 3 months before screening, inability to abstain during the study, or positive alcohol breath test (>0 mg/100 mL).
21. Excessive consumption of tea, coffee, or other caffeinated beverages (more than 8 cups/day; 1 cup = 250 mL) within 3 months prior to screening, or consumption of any caffeine within 24 hours before dosing, or unwillingness to abstain from caffeine during the study.
22. Consumption of foods or beverages that may affect drug metabolism (e.g., dragon fruit, mango, grapefruit, pomelo, orange) within 2 days before first dose, or unwillingness to avoid such items during the study.
23. Special dietary requirements that prevent adherence to standardized meals.
24. Positive pregnancy test at screening, breastfeeding, or fertile women who had unprotected intercourse within 30 days prior to screening.
25. History of needle phobia, blood phobia, or intolerance to venipuncture.
26. Vaccination within 14 days prior to screening or planned vaccination during the study.
27. Clinically significant abnormalities on physical examination, ECG, labs (CBC, urinalysis, biochemistry, coagulation, fasting C-peptide), abdominal ultrasound, or chest X-ray (PA view), as assessed by the investigator.
28. Vital signs outside the acceptable range at screening and still abnormal upon repeat measurement.
29. Any other condition that the investigator deems makes the subject unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Repaglinide | 1h before dosing, 0.25 h、0.5 h、1 h、1.5 h、2 h、3 h、4 h、6 h、8 h、12 h and 24 h post dosing
Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Rosuvastatin | 1h before dosing, 0.5 h、1 h、2 h、3 h、4 h、6 h、8 h、10 h、12 h、16 h、24 h、48 h、72 h、96 h and 120 h post dosing
Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Digoxin | 1h before dosing, 0.5 h、1 h、2 h、3 h、4 h、6 h、8 h、10 h、12 h、16 h、24 h、48 h、72 h、96 h and 120 h post dosing
Maximum Observed Concentration (Cmax) of Repaglinide | 1h before dosing, 0.25 h、0.5 h、1 h、1.5 h、2 h、3 h、4 h、6 h、8 h、12 h and 24 h post dosing
Maximum Observed Concentration of Rosuvastatin | 1h before dosing, 0.5 h、1 h、2 h、3 h、4 h、6 h、8 h、10 h、12 h、16 h、24 h、48 h、72 h、96 h and 120 h post dosing
Maximum Observed Concentration (Cmax) of Digoxin | 1h before dosing, 0.5 h、1 h、2 h、3 h、4 h、6 h、8 h、10 h、12 h、16 h、24 h、48 h、72 h、96 h and 120 h post dosing

SECONDARY OUTCOMES:
Safety of VCT220 | From day 0 to day 78
  Adverse events [TEAEs, SAEs], dose interruption, or discontinuation, vital signs (heart rate [beats/min], and changes in laboratory parameters (chemistry, hematology, urinalysis, coagulation).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No